CLINICAL TRIAL: NCT07385274
Title: Evaluation of Carotid Doppler Ultrasonography Parameters for Predicting Post-Induction Hypotension in Patients Undergoing Gynecologic Oncology Surgery: A Prospective Observational Study
Brief Title: Carotid Doppler Parameters and Post-Induction Hypotension
Acronym: CDUS-PIH
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: 1-25-1378
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Post-induction Hypotension (PIH); Gynecologic Oncology Patient; Ultrasonography, Doppler
Keywords: Corrected Flow Time; Peak Systolic Velocity; Ultrasonography, Doppler; carotid arteries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologic Oncology Surgery Cohort: Prospective observational single-center cohort of adult patients undergoing elective gynecologic oncology surgery under general anesthesia. Pre-induction carotid Doppler ultrasonography parameters were recorded to evaluate the prediction of post-induction hypotension. Baseline comorbidity burden and frailty status were assessed using the Charlson Comorbidity Index and Clinical Frailty Scale. No study-specific interventions were performed.
  Interventions: Other: pre- induction carotid doppler ultrasonography

INTERVENTIONS:
Other: pre- induction carotid doppler ultrasonography — patients undergo non-invasive carotid doppler ultrasonography

SUMMARY:
Post-induction hypotension is a common complication following the induction of general anesthesia and is associated with adverse postoperative outcomes. Patients undergoing gynecologic oncology surgery represent a particularly vulnerable population due to advanced age, high comorbidity burden, and increased frailty, which may predispose them to perioperative hemodynamic instability.

This prospective observational study aims to evaluate whether carotid Doppler ultrasonography parameters, including corrected flow time and other flow-related indices, can predict the occurrence of post-induction hypotension specifically in patients undergoing gynecologic oncology surgery.

Adult patients scheduled for elective gynecologic oncology surgery under general anesthesia will undergo pre-induction carotid Doppler ultrasonography as part of routine perioperative assessment. Baseline clinical characteristics, including the Charlson Comorbidity Index and Clinical Frailty Scale, will be recorded for each participant. Hemodynamic parameters will be recorded following anesthetic induction, and the development of post-induction hypotension will be assessed.

The findings of this study may help identify high-risk patients within the gynecologic oncology population and support the use of non-invasive carotid Doppler measurements, comorbidity burden, and frailty assessment for perioperative risk stratification in this specific surgical group.

DETAILED DESCRIPTION:
Post-induction hypotension (PIH) frequently occurs after the induction of general anesthesia and has been associated with increased perioperative morbidity, including myocardial injury, acute kidney injury, and prolonged hospital stay. Patients undergoing gynecologic oncology surgery constitute a high-risk population due to malignancy-related physiological changes, advanced age, multiple comorbidities, and increased frailty. Despite this elevated risk, data focusing specifically on predictors of PIH in the gynecologic oncology population remain limited.

Carotid Doppler ultrasonography provides real-time information about cardiac output surrogates and preload responsiveness through parameters such as corrected flow time and peak systolic velocity. These measurements may offer a practical, non-invasive method for assessing hemodynamic reserve before anesthetic induction, particularly in high-risk oncologic surgical populations.

This prospective observational study includes adult patients undergoing elective gynecologic oncology surgery under general anesthesia. Pre-induction carotid Doppler ultrasonography will be performed to obtain flow-related parameters. Baseline patient characteristics will be documented, with particular emphasis on comorbidity burden assessed using the Charlson Comorbidity Index and functional vulnerability evaluated using the Clinical Frailty Scale.

Standard anesthetic induction will be conducted according to routine clinical practice. Blood pressure measurements will be recorded before and after induction, and post-induction hypotension will be defined according to predefined criteria.

The primary objective of the study is to evaluate the association between carotid Doppler ultrasonography parameters and the development of post-induction hypotension in the gynecologic oncology population. Secondary objectives include assessment of the relationships between comorbidity burden, frailty status, Doppler-derived indices, and perioperative hemodynamic outcomes within this specific patient group.

The results of this study may contribute to improved perioperative risk assessment and support the integration of carotid Doppler ultrasonography, comorbidity indices, and frailty evaluation into routine anesthetic practice for patients undergoing gynecologic oncology surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older
* Scheduled for elective gynecologic oncology surgery under general anesthesia
* Planned standard anesthetic induction
* Ability to provide written informed consent

Exclusion Criteria:

* Refusal to participate in the study
* Inability to obtain informed consent, including patients with dementia
* Emergency surgery
* American Society of Anesthesiologists (ASA) physical status IV or higher
* Cardiac rhythm other than sinus rhythm
* Autonomic nervous system disorders
* Atrial fibrillation with rapid ventricular response
* Pregnancy
* Sepsis or septic shock
* Significant valvular heart disease or peripheral vascular disease
* Anticipated difficult ventilation and/or difficult intubation
* Left ventricular ejection fraction <40%
* Severe aortic valve stenosis
* Morbid obesity (body mass index >40 kg/m²)
* Presence of implanted cardiac pacemaker or implantable cardioverter-defibrillator
* Chronic beta-blocker therapy
* Baseline mean arterial pressure <65 mmHg at admission
* Baseline systolic arterial blood pressure >190 mmHg or diastolic arterial blood pressure >110 mmHg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult female patients aged 18 years or older undergoing elective gynecologic oncology surgery under general anesthesia. All participants are evaluated prospectively in a single-center setting. Pre-induction carotid Doppler ultrasonography is performed as part of the perioperative assessment. Baseline comorbidity burden and frailty status are assessed using the Charlson Comorbidity Index and Clinical Frailty Scale. Patients meeting predefined inclusion and exclusion criteria are enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of Post-Induction Hypotension | Within the first 20 minutes after induction of general anesthesia
  Post-induction hypotension defined as a mean arterial pressure <65 mmHg within the early post-induction period following induction of general anesthesia.

SECONDARY OUTCOMES:
Corrected Flow Time Measured by Carotid Doppler Ultrasonography | Pre-induction assessment
  Corrected flow time measured by pre-induction carotid Doppler ultrasonography and its association with post-induction hypotension.
Delta Peak Systolic Velocity Measured by Carotid Doppler Ultrasonography | Pre-induction assessment
  Delta Peak systolic velocity measured by pre-induction carotid Doppler ultrasonography and its association with post-induction hypotension.
Carotid Flow Volume Measured by Doppler Ultrasonography | Pre-induction assessment
  Carotid flow volume obtained from pre-induction Doppler ultrasonography and its relationship with the development of post-induction hypotension.
Acceleration Index Measured by Carotid Doppler Ultrasonography | Pre-induction assessment
  Acceleration index derived from pre-induction carotid Doppler ultrasonography and its association with post-induction hypotension.
Acceleration Time Measured by Carotid Doppler Ultrasonography | Pre-induction assessment
  Acceleration time measured by pre-induction carotid Doppler ultrasonography and its association with post-induction hypotension.

CONTACTS AND LOCATIONS:
Overall Officials: EMINE MUGE GOKSOY, MD, Principal Investigator — Ankara Bilkent City Hospital, University of Health Sciences, Ankara, Turkey
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to local ethical restrictions and institutional policies regarding data privacy and confidentiality.